CLINICAL TRIAL: NCT04545762
Title: A Phase 1 Clinical Trial of Anti-CD19 Chimeric Antigen Receptor T Cells for Treatment of Relapsed or Refractory Non-Hodgkin Lymphoma
Brief Title: Anti-CD19 Chimeric Antigen Receptor T Cells for Treatment of Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: C. Babis Andreadis (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor-Investigator, C. Babis Andreadis, Professor of Clinical Medicine, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19703; NCI-2020-06711 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2020-08-31; First posted 2020-09-11 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-08

CONDITIONS: Refractory Non-Hodgkin Lymphoma; Burkitt Lymphoma; Mantle Cell Lymphoma; Follicular Lymphoma; Lymphoplasmacytic Lymphoma; Primary Mediastinal Large B Cell Lymphoma; Diffuse Large B Cell Lymphoma; Small Lymphocytic Lymphoma; Transformed Lymphoma; Non-Hodgkin Lymphoma
Keywords: CAR-T Therapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Immunotherapy, Adoptive; Therapeutics; Automobiles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CLOSED TO ENROLLMENT: Dose escalation (CART-T Therapy) (Experimental): Participants will undergo Apheresis (1 day) to collect autologous lymphocytes/ mononuclear cells as per University of California, San Francisco (UCSF) institutional practices. CAR-T cell manufacturing (estimated ~13-14 days), during which participants will receive a lymphodepleting regimen of immunosuppressive chemotherapy (Cyclophosphamide 300 mg/m2/IV and fludarabine 30 mg/m2 /IV) followed by the infusion of CAR-T cells at an initial dose of 5 x 10^5 cells/kg, targeting CD19 over 5-30 minutes. Participants will be followed up 30 days after infusion, for up to 12 months, if the participant in continued remission, and for survival up to 15 years.
- Dose Expansion: Burkitt, Marginal Zone, or Waldenström Macroglobulinemia ONLY (CAR-T Therapy) (Experimental): Participants with Burkitt lymphoma, or Marginal Zone Lymphoma (MZL) and Waldenström Macroglobulinemia (WM) will undergo Apheresis (1 day) to collect autologous lymphocytes/ mononuclear cells as per University of California, San Francisco (UCSF) institutional practices. CAR-T cell manufacturing (estimated ~13-14 days), during which participants will receive a lymphodepleting regimen of immunosuppressive chemotherapy (Cyclophosphamide 300 mg/m2/IV and fludarabine 30 mg/m2 /IV) followed by the infusion of the maximum tolerated dose of CAR-T cells established in the dose escalation phase, targeting CD19 over 5-30 minutes. Participants will be followed up 30 days after infusion, for up to 12 months, if the participant in continued remission, and for survival up to 15 years.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: anti-CD19 CAR-T cells

INTERVENTIONS:
Drug: Fludarabine — Given intravenously (IV)
  Other Names: Fludarabine 30mg/m2; Fludara
  Arms: Dose Expansion: Burkitt, Marginal Zone, or Waldenström Macroglobulinemia ONLY (CAR-T Therapy)
Drug: Cyclophosphamide — Given intravenously (IV)
  Other Names: Cyclophosphamide 300mg/m2; Cytoxan; Endoxan; Neosar; Procytox; Revimmune; Cycloblastin
  Arms: Dose Expansion: Burkitt, Marginal Zone, or Waldenström Macroglobulinemia ONLY (CAR-T Therapy)
Biological: anti-CD19 CAR-T cells — Single infusion
  Other Names: CD19-directed Chimeric Antigen Receptor T-Cell (CAR T-cell) therapy; CD19-directed chimeric antigen receptor (CAR) T-cell therapy
  Arms: Dose Expansion: Burkitt, Marginal Zone, or Waldenström Macroglobulinemia ONLY (CAR-T Therapy)

SUMMARY:
This study will assess safety and feasibility of infusing genetically modified autologous T cells transduced to express a chimeric antigen receptor targeting the B cell surface antigen Cluster of Differentiation 19 (CD19).

DETAILED DESCRIPTION:
This is an open-label, pilot, phase 1 study to determine the safety profile of anti-CD19 CAR-T cell infusion in participants with R/R B-cell NHL.

PRIMARY OBJECTIVES

1. To evaluate the safety of administering chimeric antigen receptor T cells targeting CD-19 to patients with relapsed or refractory CD19+ B-cell non-Hodgkin lymphoma (NHL).
2. To determine the recommended phase 2 dose (RP2D) for this cellular therapy.

SECONDARY OBJECTIVES

1. To assess the safety and toxicity of cell collection and infusion of CAR-T cells targeting CD19 in patients with relapsed or refractory CD19+ B cell NHL.
2. To describe the efficacy of chimeric antigen receptor T cells targeting CD-19 in patients with relapsed or refractory CD19+ B cell NHL.
3. To evaluate the feasibility of CD19 CAR T cell manufacturing for patients with relapsed or refractory CD19+ B cell NHL of local manufacturing and ability to produce adequate quantities of vector positive T-cells.

OUTLINE

Participants will be enrolled to either the dose escalation or dose expansion cohorts.

Dose Escalation: CLOSED TO ENROLLMENT

Dose Expansion: The dose expansion phase of the study will be limited to two disease-specific cohorts:

* Cohort B: Participants with Burkitt lymphoma (B).
* Cohort M/W: Participants with Marginal Zone Lymphoma (MZL) and Waldenström Macroglobulinemia (WM).

Participants will receive an infusion of Anti-CD19 CAR-T cells during the main study and will be followed for 12 months before being transferred into long term follow-up during years 1 to 15.

ELIGIBILITY:
THE DOSE ESCALATION COHORT IS CLOSED TO FURTHER ENROLLMENT.

Inclusion Criteria:

Dose expansion Cohorts:

Cohort B (Burkitt):

1. Participants must have a diagnosis of relapsed or refractory Burkitt Lymphoma

   * Participants with Burkitt lymphoma must have relapsed or failed to respond to at least 1 prior line of multiagent chemoimmunotherapy with prior exposure to both an anti-CD20 antibody agent and an anthracycline.
   * No significant circulating disease, defined as an elevated total lymphocyte count above the upper limit of normal (ULN) due to the presence of malignant cells.
2. Participants must have measurable disease as defined below:

   * Participants with Burkitt Lymphoma must have Positron Emission Tomography (PET)-positive disease according to "Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification"

Cohort M/W (Marginal/Waldenström):

1. Participants must have a diagnosis of relapsed or refractory Marginal Zone Lymphoma (MZL), or Lymphoplasmacytic Lymphoma (LPL)/Waldenström Macroglobulinemia (WM):

   o Participants with indolent lymphomas (nodal or extranodal marginal zone lymphoma, and lymphoplasmacytic lymphoma) must have relapsed after or have been refractory to ≥ 2 prior lines of multi-agent chemoimmunotherapy including prior exposure to an anti-CD20 antibody and an alkylating agent.
2. Participants must have measurable disease as defined below:

   o Participants with Marginal Zone Lymphoma or Lymphoplasmacytic Lymphoma/Waldenström Macroglobulinemia: must either have PET-positive disease according to "Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification" or serum monoclonal immunoglobulin M (IgM) paraprotein > 0.5 g/dL.
3. Participants with indolent lymphoma (Marginal Zone Lymphoma or Lymphoplasmacytic Lymphoma/Waldenström Macroglobulinemia) must have symptomatic disease necessitating systemic treatment.

In addition, all participants must meet the following criteria:

1. CD19-positive by either immunohistochemistry or flow cytometry analysis on any biopsy. If prior anti-CD19 therapy has been administered, CD19-positivity has to be re-established on the most recent biopsy.
2. Age ≥18 years at the time of consent.
3. Absolute lymphocyte count > 100/UL.
4. Eastern Cooperative Oncology Group (ECOG) performance status < 2.
5. Adequate organ function, defined as:

   1. Adequate bone marrow function for apheresis and lymphodepleting chemotherapy
   2. Hemoglobin >8 gm/dl (transfusions allowed)
   3. Platelets >50,000/uL (transfusions allowed)
   4. Absolute Neutrophil Count (ANC) > 500/uL
   5. alanine aminotransferase (ALT)/aspartate aminotransferase (AST) < 3 x institutional upper limit of normal (ULN) and Total bilirubin < 1.5 mg/dl x institutional ULN, except with Gilbert's syndrome
   6. Serum Creatinine < 2 x the institutional ULN
   7. Adequate cardiac function, defined as left ventricular ejection fraction (LVEF) > 40% as assessed by echocardiogram or multiple uptake gated acquisition (MUGA) within 3 months of screening. Repeat testing may occur at Investigator's discretion.
6. Adequate vascular access for leukapheresis procedure (either peripheral line or surgically placed line).
7. Women of childbearing potential (defined as all women physiologically capable of becoming pregnant) must have a negative serum or urine pregnancy test AND agree to use highly effective methods of contraception for 1 year after the last dose of anti-CD19 CAR-T cells.
8. Males who have partners of childbearing potential must agree to use an effective barrier contraceptive method.
9. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Autologous transplant within 6 weeks of planned CAR-T cell infusion.
2. Recipient of prior CAR-T cell therapy targeting CD19 outside of this protocol.
3. Active other malignancy, other than non-melanoma skin cancer, carcinoma in situ (e.g., cervix, bladder, or breast).
4. Human immunodeficiency virus (HIV) seropositivity.
5. Serologic status reflecting active hepatitis B or C infection. Participants that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive participants will be excluded.)
6. Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant or breastfeeding women are excluded from this study because CAR-T cell therapy may be associated with the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with CAR-T cells, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study. NOTE: Women of childbearing potential must have a negative serum or urine pregnancy test.
8. Participants with history of clinically relevant central nervous system (CNS) pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia and Parkinson's disease.
9. History of autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus) with requirement of immunosuppressive medication within 6 months.
10. Body weight <40 kilograms(kg).

Eligibility for Infusion of Investigational Product:

Participants will undergo an evaluation of eligibility on day 1 prior to infusion of anti-CD19 CAR-T cell product. This eligibility criterion will include the inclusion and exclusion criteria required for enrollment with the following exceptions and additions:

1. No significant laboratory abnormalities. Laboratory result abnormalities that are considered not clinically significant by the principal investigator AND are not the result of a demonstrated active infection or an active central nervous system condition.
2. ECOG performance status < 2
3. No evidence of uncontrolled intercurrent illness including, but not limited to ongoing or active infection, inflammatory response, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities or psychiatric illness/social situations.
4. No new neurologic symptoms suggestive of an active central nervous system condition, or uncontrolled CNS involvement by lymphoma.
5. No corticosteroid use within 7 days prior to infusion (with exception of agents used for prevention of emesis during lymphodepletive chemotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with treatment-emergent adverse events (AEs) | From initiation of study treatment to 12 months following CAR-T infusion, approximately 15 months
  Participants treated with conforming product who received the target doses of anti-CD19 CAR-T infusion will be included in the analysis. Proportion of participants with treatment-emergent adverse events of CAR-T in B-cell NHL, as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5.0), revised Cytokine Release Syndrome (CRS) grading criteria, and American Society for Transplantation and Cellular Therapy (ASTCT) immune effector cell (IEC) -associated neurotoxicity syndrome (ICANS) Consensus Grading for Adults (for neurotoxicity grading).
Proportion of participants who experience a dose-limiting toxicity (DLT) (Dose escalation) | From initiation of study treatment to 30 days following CAR-T infusion
  A DLT includes AEs graded according to CTCAE version 5.0, with the exceptions of CRS and neurotoxicity, which are graded using CRS and ICANS criteria. DLTs must 1) be suspected to be secondary to CAR-T cell infusion, 2) occur during the first 30 days after infusion and 3) meet the following criteria: 1. Grade 3 or 4 non-hematologic toxicities of any duration, with following exceptions: Grade 3 laboratory abnormalities without associated symptomatology or clinical consequence that resolve in < 7 days; AEs associated with Grade <= 2 CRS; Toxicities associated with Grade 3 CRS (except cardiac or pulmonary organ toxicity) that improves to grade <= 2 within 3 days of intervention; isolated renal or hepatic grade 3 organ toxicity that does not resolve within 7 days; Laboratory abnormalities compatible with tumor lysis syndrome; Grade 4 hematological toxicity that persists at grade >= 3 despite maximum supportive care for >21 days.

SECONDARY OUTCOMES:
Proportion of participants with CAR-T infusion related adverse events (Dose Escalation) | From initiation of CD19 CAR T-cell manufacturing to end of infusion, approximately 18 days
  The proportion of participants with adverse events related to the collection and infusion of CAR-T cells targeting CD19 will be reported.
Proportion of participants with delayed infusion due to study-related adverse events | From T-cell collection to end of infusion, approximately 18 days
  The proportion of participants who have their infusion delayed due to and AE will be reported.
Overall Response Rate (ORR) | From initiation of study treatment to 12 months after getting CAR-T infusion, approximately 15 months
  Overall response rates will be reported as proportions of participants by arm. The 2014 Lugano Response for Malignant Lymphoma criteria will be to determine response: Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Relapse and Progression (PD). For the Waldenstrom's Macroglobulinemia cohort, the 11th International Workshop on Waldenstrom's Macroglobulinemia (IWWM-11) response criteria will be used to determine response: CR, very good partial response (VGPR), PR, minor response (MR), SD, and PD.
Complete Response Rate | From initiation of study treatment to 12 months after getting CAR-T infusion, approximately 15 months
  Complete response rates will be reported as will be reported as proportions of participants by arm.
Partial Response Rate | From initiation of study treatment to 12 months after getting CAR-T infusion, approximately 15 months
  Partial response rates will be reported as will be reported as proportions of participants by arm.
Median duration of response | From initiation of study treatment to 12 months after getting CAR-T infusion, approximately 15 months
  For participants who have been documented to be responders under the 2014 Lugano criteria or the IWWM-11 criteria, and defined as the median time from the documented beginning of response (CR or PR) to the time of relapse.
Median Progression-free Survival (PFS) | From initiation of study treatment to 12 months after getting CAR-T infusion, approximately 15 months
  PFS is defined as the median time from entry onto study until a diagnosis of lymphoma progression or death from any cause at 12 months after receiving CAR-T infusion.
Median Overall Survival | Up to 15 years
  Defined as the median time from entry onto study until death from any cause
Proportion of participants for whom CD19 CAR T-cell therapy is manufactured | From initiation of CD19 CAR T-cell manufacturing to end of infusion, approximately 18 days
  The proportion of participants for whom CD19 CAR T-cell therapy is adequately manufactured and meets pre-specified release criteria.
Proportion of participants who complete study treatment | From initiation of CD19 CAR T-cell manufacturing to end of infusion, approximately 18 days
  Feasibility will be assessed by the proportion of participants who are able to complete the study regimen and receive infusion of CAR-T therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Ho, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338